CLINICAL TRIAL: NCT03271710
Title: A Single-Arm, Multicenter Study for the Lower Extremities Using the Vanguard IEP Peripheral Balloon Angioplasty System With Integrated Embolic Protection
Brief Title: Study to Evaluate the Lower Extremity Intervention With Integrated Embolic Protection Using the Vanguard IEP System
Acronym: ENTRAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Contego Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSP1121
Record Dates: First submitted 2017-04-26; First posted 2017-09-05 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Peripheral Arterial Disease; Intermittent Claudication; Atherosclerosis of Femoral Artery
Keywords: Distal embolization; Percutaneous transluminal angioplasty; Integrated embolic protection
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication | interventions — Angioplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Peripheral balloon angioplasty (Experimental): Peripheral vascular percutaneous transluminal angioplasty (PTA) and capture and removal of embolic material during angioplasty for the femoral, iliac, popliteal and profunda arteries with the Vanguard IEP Peripheral Balloon Angioplasty System with Integrated Embolic Protection
  Interventions: Device: peripheral balloon angioplasty

INTERVENTIONS:
Device: peripheral balloon angioplasty — Percutaneous transluminal angioplasty (PTA) of the lower extremities
  Other Names: percutaneous transluminal angioplasty (PTA)

SUMMARY:
The ENTRAP Study is a prospective, multi-center, non-randomized, single-arm, study with follow-up to 30 days to determine the acute safety, acute device performance and clinical performance of the Vanguard IEP Peripheral Balloon Angioplasty System with Integrated Embolic Protection. The Vanguard IEP Peripheral Balloon Angioplasty System with Integrated Embolic Protection is indicated for peripheral vascular percutaneous transluminal angioplasty (PTA) and capture and removal of embolic material during angioplasty for the femoral, iliac, popliteal and profunda arteries.

DETAILED DESCRIPTION:
The ENTRAP Study is a prospective, multi-center, non-randomized, single-arm, study with follow-up to 30 days to determine the acute safety, acute device performance and clinical performance of the Vanguard IEP Peripheral Balloon Angioplasty System with Integrated Embolic Protection. The Vanguard IEP Peripheral Balloon Angioplasty System with Integrated Embolic Protection is indicated for peripheral vascular percutaneous transluminal angioplasty (PTA) and capture and removal of embolic material during angioplasty for the femoral, iliac, popliteal and profunda arteries.

The Vanguard System has been designed to revascularize iliac and femoro-popliteal PAD while protecting against embolization at the same time. It is the first system in which the embolic protection filter is coupled on the same catheter as the angioplasty balloon for use in the lower extremities. Up to 130 patients will be enrolled into this study and followed for 30 days after post-procedure. Adult patients with lifestyle-limiting claudication or rest pain (Rutherford categories 2 to 3) who meet all eligibility criteria will be approached for participation in the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients ≥18 years old.
2. Subject has clinically significant symptomatic leg ischemia requiring treatment.
3. Subject has a Rutherford category of 2 - 3.
4. Target lesion in the superficial femoral artery (SFA), common femoral artery, p1 segment of popliteal artery, common iliac artery and external iliac artery (cross-over access only), and profunda femoris arteries.
5. Target lesion stenosis >50% by investigator's visual estimate.
6. Vessel diameter between 4.0 mm and 8.0 mm at the site of the target lesion.
7. Total target lesion length ≤ 18 cm, and may include a chronic total occlusion ≤ 10 cm.
8. If target lesion is restenotic, the prior PTA must be > 30 days prior to enrollment.
9. If the guide wire traverses the lesion subintimally, it must enter the true lumen distal to the lesion without the use of a reentry device.
10. Distal vessel diameter at the site of filter deployment of 4.0 mm to 8.0 mm with sufficient landing zone required for the successful deployment of the integrated embolic protection filter.
11. Patent popliteal and infrapopliteal arteries; I.e. single vessel runoff or better with at least one of three vessels patient (<50% stenosis) to the ankle or foot.
12. The patient (or legally authorized representative) is willing to provide written informed consent and to comply with all study requirements.

Exclusion Criteria:

1. Subjects who have undergone prior vascular surgery of the target artery to treat atherosclerotic disease.
2. History of major amputation in the same limb as the target lesion.
3. Woman who is pregnant or nursing.
4. Subject has Rutherford category of 4- 6.
5. Target lesion(s) within native or synthetic vessel grafts.
6. Use of atherectomy as an adjunctive therapy during the index procedure in the target lesion or target vessel.
7. Any major (e.g. cardiac, peripheral, abdominal) intervention, including in the contralateral lim planned within 30 days post index procedure.
8. Presence of other hemodynamically significant outflow lesion in the target limb requiring intervention within 30 days of enrollment.
9. Subject has significant inflow disease which cannot be treated prior to target lesion treatment.
10. Presence of aneurysm in the target vessel.
11. Acute limb occlusion due to thrombotic occlusion of the target limb.
12. In-stent restenosis of target lesion.
13. Severe calcification that renders the target lesion lesion resistant to angioplasty.
14. Visible acute thrombus in the target lesion
15. Intolerance to antiplatelet, anticoagulant or thrombolytic therapy medications that would be administered during the trial.
16. Known hypersensitivity to contrast media that cannot be adequately premedicated.
17. Known hypersensitivity to nickel and/or titanium.
18. Acute Myocardial Infarction within 30 days prior to the index procedure.
19. Subject has a known coagulopathy or bleeding diathesis, or INR <1.5.
20. Platelet count <100,000 mm3/L or >700,000 mm3/L
21. Concomitant renal failure with a serum creatinine > 2.5 mg/dL or receiving dialysis.
22. Patient is currently participating in an interventional study, investigational drug or device study that has not completed the primary endpoint, that may potentially confound the results of this trial or that would limit the subject's compliance with the follow-up requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Freedom from MAE, defined as death, amputation and target vessel revascularization (TVR) | 30 days
  Primary safety endpoint
Procedural success | 24 hours or at discharge.
  Defined as <50% residual stenosis without MAE (death, amputation or TVR)

SECONDARY OUTCOMES:
Technical Success | Index procedure
  Technical success of the investigational device using questionnaire
Ankle-Brachial Index (ABI) | Baseline, discharge and 30 days
  Change in Ankle-Brachial Index from baseline, discharge and 30 days
Rutherford-Becker | 30 days
  Rutherford-Becker improvement greater than or equal to 1

OTHER OUTCOMES:
Histomorphometric analysis of embolic protection filter content | Day 0. Filter collected at end of index procedure.
  Histomorphometric analysis of embolic protection filter content

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Zeller, Prof., Principal Investigator — Universitäts-Herzzentrum Freiburg
Locations (9):
- Belgium (4):
  - OLV Hospital Aalst, Aalst
  - Imelda Hospital / Vascular Science Research Center, Bonheiden
  - AZ Sint Blasius, Dendermonde
  - RZ Heilig Hart Hospital, Tienen
- Germany (5):
  - Interventional Cardiology and Vascular Medicine, Department of Angiology, Universitäts-Herzzentrum Freiburg, Bad Krozingen
  - Sankt Gertrauden-Krankenhaus, Berlin
  - Daikonissenkrankenhaus Flensburg, Flensburg
  - MVZ/Prof. Mathey Prof. Schofer Clinic, Hamburg
  - Universitätsklinikum Leipzig, Leipzig

IPD SHARING:
Plan to Share IPD: No
Site specific individual participant data is available to each research site via export from EDC.